CLINICAL TRIAL: NCT02020031
Title: Regional Prophylactic Vancomycin in Revision Total Knee Replacement
Acronym: VIDACARE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Vidacare Corporation (Industry)
Responsible Party: Principal Investigator, Mark J. Spangehl, M.D., PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-004988
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Results first posted 2016-11-25 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-10

CONDITIONS: Arthropathy of Knee Joint
Keywords: Revision knee joint
MeSH Terms: interventions — Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vancomycin 500mg intraosseous (Experimental): Vancomycin 500mg is given via intraosseous regional administration (IORA) into a proximal tibial cannula, after tourniquet inflation and immediately prior to skin incision.
  Interventions: Drug: Vancomycin
- Vancomycin 1g IV (Active Comparator): Vancomycin 1g is administered via forearm vein, given over a one-hour infusion, timed to finish approximately 30 minutes prior to tourniquet inflation.
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Vancomycin
  Other Names: Vancocin

SUMMARY:
The purpose of this study is to determine whether or not giving a lower dose of antibiotics (Vancomycin) in the area where it is needed (the knee joint) is more effective at preventing infection than the current standard dose which is given intravenously (IV) through a wrist vein.

DETAILED DESCRIPTION:
Patients were assigned to one of two groups by chance (like a coin toss):

* GROUP 1 - Received 500mg of vancomycin into the tibia (shin) bone of the leg being operated on.
* GROUP 2 - Received 1g of vancomycin, which is the amount normally given to patients.

For both groups, the revision knee replacement will then be carried out as normal.

OTHER ANTIBIOTICS All patients received cefazolin IV (an antibiotic used to prevent infection) prior to the beginning of surgery to ensure effective preventive antibiotics. The patient will also received 3 postoperative doses of cefazolin over a 24-hour period (4 doses in total). This is standard of care for all total knee replacement surgeries.

TISSUE SAMPLES

* Ten (10) tissue samples were taken during the surgery, consisting of both bone and fat beneath the skin. Each sample were very small, around the size of a pinhead.
* In addition, a drain sample was taken from the knee joint drain fluid to measure vancomycin concentration the morning following surgery.
* These samples were frozen and sent to a lab for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Revision total knee arthroplasty
* Informed consent given

Exclusion Criteria:

* Current treatment with IV Vancomycin within the preceding 7 days
* Previous hypersensitivity to vancomycin
* Significant cardiac or respiratory abnormality
* Contraindications to using the intraosseous vascular access system (EZ-IO)
* Sepsis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Spangehl, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled between January 2014 and April 2015 at Mayo Clinic in Arizona.
Period: Overall Study
Arm/Group | Vancomycin 500mg Intraosseous | Vancomycin 1g IV
Started | 11 | 11
Completed | 10 | 10
Not Completed | 1 | 1
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Population: Although 22 subjects were enrolled, 2 subjects were withdrawn from the study following an intra-operative decision not to proceed with a full revision. Baseline demographics are provided for the subjects who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vancomycin 500mg Intraosseous | Vancomycin 1g IV | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Full Range); unit: years] | 69.3 [43 to 83] | 67.4 [54 to 82] | 68.4 [43 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 3 | 5 | 8
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Mean Concentration of Vancomycin in Subcutaneous Fat
Description: During the procedure, subcutaneous fat samples (approximately 0.5 cm^3) were taken at regular intervals until skin closure. Vancomycin concentrations were determined by liquid chromatography coupled with tandem mass spectrometry. Times are given as minutes post surgical incision.
Time Frame: Baseline to 24 hours
Measure: Mean (Standard Deviation); unit: µg/g
Arm/Group | Vancomycin 500mg Intraosseous | Vancomycin 1g IV
Number analyzed (Participants) | 10 | 10
µg/g
  At approximately 3 minutes | 94.1 (69.0) | 3.2 (1.8)
  At approximately 30 minutes | 88.3 (131) | 5.0 (2.9)
  At approximately 50 minutes | 69.4 (50) | 4.2 (2.5)
  At approximately 115 minutes | 173 (445) | 4.7 (2.6)
  At approximately 150 minutes | 249 (639) | 4.0 (2.2)
  At approximately 180 minutes | 18.2 (11.6) | 3.6 (2.5)
Statistical Analysis 1: Comparison: Vancomycin 500mg Intraosseous vs Vancomycin 1g IV; Comparison at approximately 3 minutes, adjusted by BMI, age, and length of surgical procedure; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: Vancomycin 500mg Intraosseous vs Vancomycin 1g IV; Comparison at approximately 30 minutes, adjusted by BMI, age, and length of surgical procedure; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 3: Comparison: Vancomycin 500mg Intraosseous vs Vancomycin 1g IV; Comparison at approximately 50 minutes, adjusted by BMI, age, and length of surgical procedure; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 4: Comparison: Vancomycin 500mg Intraosseous vs Vancomycin 1g IV; Comparison at approximately 115 minutes, adjusted by BMI, age, and length of surgical procedure; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 5: Comparison: Vancomycin 500mg Intraosseous vs Vancomycin 1g IV; Comparison at approximately 150 minutes, adjusted by BMI, age, and length of surgical procedure; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 6: Comparison: Vancomycin 500mg Intraosseous vs Vancomycin 1g IV; Comparison at approximately 180 minutes, adjusted by BMI, age, and length of surgical procedure; Test type: Superiority or Other; p < 0.0001, ANOVA

2. Primary Outcome: Mean Concentration of Vancomycin in Bone Samples
Description: During the procedure, bone samples (approximately 0.5 cm^3) were taken at regular intervals were taken at regular intervals until skin closure. All bone samples were taken from the femur, distant from the tibial intraosseous injection site. Vancomycin concentrations were determined by liquid chromatography coupled with tandem mass spectrometry. Times are given as minutes post surgical incision.
Time Frame: baseline to 24 hours
Measure: Mean (Standard Deviation); unit: µg/g
Arm/Group | Vancomycin 500mg Intraosseous | Vancomycin 1g IV
Number analyzed (Participants) | 10 | 10
µg/g
  At approximately 30 minutes | 90.7 (77) | 7.9 (5.7)
  At approximately 50 minutes | 193 (191) | 8.6 (5.9)
  At approximately 115 minutes | 59.8 (63) | 5.0 (2.3)
  At approximately 145 minutes | 62.9 (62) | 7.1 (4.4)

ADVERSE EVENTS:
Arm/Group | Vancomycin 500mg Intraosseous | Vancomycin 1g IV
Serious Adverse Events (participants affected / at risk) | 4/10 | 0/10
Other Adverse Events (participants affected / at risk) | 5/10 | 3/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vancomycin 500mg Intraosseous (N=10) | Vancomycin 1g IV (N=10)
Acute renal failure with olgiurea (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute blood loss anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Intraoperative opiate overdose (Surgical and medical procedures) | 1 (1) | 0 (0) — Required postoperative infusion of Narcan
Postoperative hypoxemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Secondary to acute asthma exacerbation; pulmonary embolism ruled out.
Foot drop of left leg (Nervous system disorders) | 1 (1) | 0 (0)
Left peroneal neuropathy (Nervous system disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vancomycin 500mg Intraosseous (N=10) | Vancomycin 1g IV (N=10)
Altered mental state (Psychiatric disorders) | 1 (1) | 0 (0)
Hypotension (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Intermittent atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Hyponatremia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Procedure turned into a brief operation and not full revision (Surgical and medical procedures) | 0 (0) | 1 (1) — Patient withdrawn and study collection terminated
Pulmonary bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — With oxygen desaturation with leg swelling
Hypovolemic hyponatremia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Premature ventricular complexes (Cardiac disorders) | 0 (0) | 1 (1)
Elevated temperature post surgery (General disorders) | 2 (2) | 0 (0)
Swelling below eyes (General disorders) | 1 (1) | 0 (0) — Possibly due to intraoperative fluid volume and positioning
Replacement of thoracic pulse generator (Surgical and medical procedures) | 1 (1) | 0 (0) — Device could not be started up after patient's knee surgery. Patient has history of cervical enteropathic syndrome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes